CLINICAL TRIAL: NCT04392934
Title: The Short-term Effects of a Conservative Physiotherapy Method in Subacromial Impingement Syndrome and Its Relation to Acromion Morphology
Brief Title: Conservative Physiotherapy and Acromion Morphology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Begümhan Turhan, Assistant Professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/100
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Subacromial Impingement Syndrome; Morphologic Change
Keywords: physiotherapy; acromion morphology; subacromial impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are grouped according to their acromion type. First group is flat shape acromion group, second is hook shape group and the third one is curved shape acromion group. All groups are treated with the same physiotherapy protocol.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- flat shape acromion group (Experimental): a conservative physiotherapy protocol was applied for 4 weeks
  Interventions: Procedure: a conservative physiotherapy protocol
- curved shape acromion group (Experimental): a conservative physiotherapy protocol was applied for 4 weeks
  Interventions: Procedure: a conservative physiotherapy protocol
- hooked shape acromion group (Experimental): a conservative physiotherapy protocol was applied for 4 weeks
  Interventions: Procedure: a conservative physiotherapy protocol

INTERVENTIONS:
Procedure: a conservative physiotherapy protocol — 5 minutes of ultrasound (Business Line US 50, Medical Italia, Italy) at a frequency of 1 MHz and intensity of 1.5 watts/cm², 20 minutes of conventional TENS (BTL-5000, UK ) applied to the patients. Then Codman's exercises, shoulder wheel activity, isometric exercises, range of motion exercises, capsular stretching, scapular stabilization exercises, and muscle strengthening exercises were done by patients. After the treatment, cold pack was applied to the shoulder for 10 minutes. The modalities in the treatment program were applied for a total of 20 sessions 5 days per week.

SUMMARY:
In this study, we aimed to evaluate the short-term effects of conservative physiotherapy in the subacromial impingement syndrome (SIS) and its relation to the acromion morphology.

DETAILED DESCRIPTION:
The aim of this study is to investigate the short term effects of physiotherapy in SIS patients on pain, range of motion, muscle strength, joint position sense and functionality and its relation to the acromion shape. Fifty patients (26 female, 24 male) with SIS were evaluated in this study. Patiens were divided into 3 groups according to the their acromion morphology. A conservative physiotherapy method was applied to the patients. All patients were evaluated before and 4 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed (clinically and by MRI) with SIS by the physician, at a stage of II-III levels according to Neer's criteria, who were undergoing physiotherapy for the first time and who had not received any treatment from the shoulder region before were included in this study.

Exclusion Criteria:

* Patients who had a history of fracture in the upper extremity and, surgical operation from any part of the upper extremity, who had acute cervical disc herniation or a neuromuscular disease, receiving a medical therapy for pain relief, less than 80 % participation to sessions were excluded.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 weeks
  Pain at rest and pain at activity was measured by Visual Analog Scale (VAS). High score was determined as high level of pain. Visual analog scale (VAS) was ranging from 0 cm (no pain) to 10 cm (worst imaginable pain).
Muscle strength | 4 weeks
  Muscle strength tests for shoulder flexion, extension, abduction, adduction, internal and external rotation were done by a dynamometer (NK-500, AIPU, Anhui, China).
Range of motion | 4 weeks
  Goniometric measurements were applied by a universal goniometer to determine the range of motion in terms of flexion, extension, abduction, adduction, internal and external rotation directions.
Joint position sense | 4 weeks
  The joint position sense was evaluated by a laser pointer. During the test, 90˚ shoulder flexion and 90˚ shoulder abduction movements were evaluated. A laser pointer was fixed with a velcro 5 cm above the elbow. The patient was asked to bring the shoulder to 90˚ flexion while the patient's eyes were open and meanwhile, the measurement was made by the physiotherapist with a goniometer. The patient was asked to fix this position for 10 seconds. The projection of the laser pointer on millimeter paper was marked. The patient repeated this movement 3 times with eyes open and memorized it. The patient returned to the neutral position and closed her eyes then repeated the flexion movement 3 times and the projection of the laser pointer on millimeter paper was marked. The same procedure was performed for shoulder abduction. The deviation between the measurements was calculated.
Painful arc sign | 4 weeks
  The patient was asked to perform active shoulder abduction, and the difference between the angle at which the pain first occurred and the angle at which the pain ended was noted during this movement pattern. Measurements were made on the affected shoulder joint by a goniometer
Functionality | 4 weeks
  To assess the functional levels of the patients, the Shoulder Pain and Disability Index (SPADI) was used.

CONTACTS AND LOCATIONS:
Overall Officials: Begumhan Turhan, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)